CLINICAL TRIAL: NCT03026543
Title: A Prospective, Blinded, Randomized Clinical Trial Investigating the Effect on Postoperative Pain and Nausea, When Performing a Ventilator-piloted PRM at the End of Laparoscopic Cholecystectomy
Brief Title: Effect of Pulmonary Recruitment Maneuver (PRM) on Pain and Nausea After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Ebba Kihlstedt Pasquier, Principal Investigator, Region Östergötland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Regionostergotland
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Cholecystectomy, Laparoscopic; Ventilators, Mechanical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Pulmonary recruitment maneuver (Experimental): One minute of ventilator-piloted PRM at the end of laparoscopic cholecystectomy, intending to remove residual carbon dioxide (CO2) from the abdomen.
  Interventions: Procedure: Pulmonary Recruitment Maneuver; Procedure: Laparoscopic cholecystectomy; Device: Ventilator
- Control group (Active Comparator): Ordinary ventilation at the end of laparoscopic cholecystectomy.
  Interventions: Procedure: Laparoscopic cholecystectomy; Device: Ventilator

INTERVENTIONS:
Procedure: Pulmonary Recruitment Maneuver
  Arms: Pulmonary recruitment maneuver
Procedure: Laparoscopic cholecystectomy
Device: Ventilator

SUMMARY:
This prospective, blinded, randomized clinical trial investigates the effect on postoperative pain and nausea, when performing a ventilator-piloted PRM at the end of a laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic cholecystectomy
* American Society of Anesthesiologists (ASA) physical status classification I-II (with the exception of body mass index over 35 kg/m2)
* written consent

Exclusion Criteria:

* conversion to open surgery
* Clavien-Dindo grade ≥ II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain assessed with a numeric rating scale | 4, 12, 24, 36 and 48 hours after surgery
  A questionnaire with a numeric rating scale (NRS) is used to assess pain intensity at 4, 12, 24, 36 and 48 hours postoperatively.

SECONDARY OUTCOMES:
Change in postoperative nausea assessed with a Questionnaire | 4, 12, 24, 36 and 48 hours after surgery
  A questionnaire is used to evaluate nausea at 4, 12, 24, 36 and 48 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ebba Kihlstedt Pasquier, MD, Principal Investigator — Vrinnevi Hospital, Norrköping, Sweden; Ellen Andersson, MD, PhD, Study Chair — Vrinnevi Hospital, Norrköping, Sweden
Locations (1):
- Vrinnevi Hospital, Norrköping, Östergötland County, Sweden

REFERENCES:
- [Result] Kihlstedt Pasquier E, Andersson E. Pulmonary Recruitment Maneuver Reduces Shoulder Pain and Nausea After Laparoscopic Cholecystectomy: A Randomized Controlled Trial. World J Surg. 2021 Dec;45(12):3575-3583. doi: 10.1007/s00268-021-06262-6. Epub 2021 Sep 5. PMID 34482412